CLINICAL TRIAL: NCT02492087
Title: Prophylactic Use of Topical Tranexamic Acid to Aid Surgical Haemostasis During Caesarean Sections in Parturients With Moderate to High Risk of Bleeding
Brief Title: Topical Tranexamic Acid in Caesarean Section
Acronym: TXACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Meng-Li Lee (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor-Investigator, Dr Meng-Li Lee, Specialist Anaesthetist, Ministry of Health, Malaysia
Organization: Ministry of Health, Malaysia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NMRR-14-1034-20129
Record Dates: First submitted 2015-06-18; First posted 2015-07-08 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Haemorrhage
Keywords: topical; tranexamic acid; haemostasis; caesarean section; bleeding; postpartum hemorrhage; prophylactic
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Tranexamic Acid; Saline Solution; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (TXA) Group (Active Comparator): Subjects in the TXA group will receive the topical tranexamic acid solution which will be administered intra-operatively, during the caesarean section on the surgical wound and into the intrauterine cavity after the delivery of the baby and the placenta. 60mls of the solution will be applied topically to the placental bed as identified by the surgeon carrying out the surgery by spraying the study solution using a syringe into the uterine cavity. Another 30mls of the solution will be applied to the open incision wound. The surgeon will then proceed to close the first layer of the uterus in the usual manner. The remaining 30mls of the study drug solution is then applied topically on the closed incision wound
  Interventions: Drug: Topical tranexamic acid
- Control Group (Sham Comparator): Subjects in the Control group will receive topical normal saline solution which will be administered intra-operatively in the same manner as described for the TXA group.
  Interventions: Drug: Normal saline 0.9%

INTERVENTIONS:
Drug: Topical tranexamic acid — Topical tranexamic acid 2g diluted with normal saline 0.9% to a volume of 120mls solution (Concentration 16.7mg/ml)
  Other Names: TXA group
  Arms: Tranexamic acid (TXA) Group
Drug: Normal saline 0.9% — Sterile Normal saline 0.9% 120mls solution
  Other Names: Control group
  Arms: Control Group

SUMMARY:
The objective of this study is to investigate whether topical application of tranexamic acid into the uterine cavity and the surgical site intra-operatively can reduce blood loss and provide better surgical haemostasis in parturients with moderate to high risk for bleeding undergoing caesarean deliveries.

DETAILED DESCRIPTION:
1.1 BACKGROUND

Maternal haemorrhage is a significant cause of maternal mortality and morbidity worldwide. The incidence of postpartum haemorrhage (PPH) with blood loss in excess of 1000ml is estimated to affect 10.5% of live births globally. This translate to a staggering number of 14 million women in the reproductive age group who suffers from complications of severe blood loss during childbirth every year. While the case fatality rate is low at around 1%, non-fatal health outcomes as a result of PPH remains unknown and this is further compounded by considerable variability in patients tolerance towards blood loss.

Certainly, not all parturients experience similar risks for bleeding during their pregnancy. However, it is important to consider that even small amounts of blood loss may have a detrimental effect on maternal health especially in parturients with preexisting medical conditions like anaemia or cardiac disease. Measures aimed at addressing this global problem need to be given top priority in line with the United Nations Fifth Millennium Developmental Goal to improve maternal health and to reduce maternal mortality ratio by 75% by the year 2015.

Parturients undergoing caesarean section experience more blood loss compared to their counterparts who deliver vaginally. Recent studies reported average blood loss of 254ml to 304ml for vaginal deliveries and 500ml to 592ml for caesarean deliveries. Identifying the risks and causes of PPH and recognising that PPH is a significant contributor to maternal mortality and morbidity is important to encourage efforts for early identification of parturients at risk of bleeding. However, despite the advances in modern obstetrics, PPH remains a significant problem not only in the developing world but also in countries with high resources and better medical facilities and presumably where more efficient protocols for management of PPH are in existence.Obviously, this indicate the need to explore newer methods for more effective prevention and treatment of PPH in the quest to improve maternal health.

1.2 INVESTIGATIONAL AGENT AND MECHANISM OF ACTION

Tranexamic acid, a tissue plasmin and plasminogen inhibitor, is a widely used drug which has showed benefit in reducing blood loss in various surgical specialties. It acts by reversible blocking the lysine binding sites of plasminogen and preventing its activation to plasmin. This inhibits the fibrinolytic process and prevent breakdown of polymerized fibrin, which is necessary for the blood clot to form.

In this study, the investigators proposed the use of prophylactic administration of topical tranexamic acid given intra-operatively to parturients with moderate to high risk of bleeding undergoing caesarean sections, as part of the blood conservation strategy to aid surgical haemostasis and reduce blood loss. This relatively simple and easy to administer route of tranexamic acid is postulated to inhibit the local fibrinolytic process at the site of tissue injury. Bleeding in caesarean section can occur from the surgical incision site, from vessel injuries and from the placental separation site in the uterus. The investigators postulate that by applying tranexamic acid locally at these sites, a reduction in blood loss can be achieved and thus help prevent the occurrence of PPH and reduce the risk for blood transfusion.

1.3 CLINICAL DATA TO DATE

A few systematic reviews have been conducted in the past and the use of systemic and topical tranexamic acid in trauma, cardiac, spine and arthroplasty surgeries have mostly shown favourable outcomes. However, the evidence for use of tranexamic acid in obstetrics patients remains limited. A Cochrane review in 2010 of tranexamic acid for preventing PPH confirms the poor state of evidence in this area. The EXADELI (EXAcyl in the treatment of DELIvery haemorrhage) study shows reduction in median blood loss after 6 hours in the treatment group who received a high dose of tranexamic acid (4g in 1h followed by 1g/h) in women who develop PPH of more than 800ml within 2 hours of vaginal delivery. There is also a large international multi-centred randomised controlled trial currently in progress to investigate the use of systemic tranexamic acid in treating PPH in both vaginal and caesarean delivery (WOMAN trial) and its outcome is awaited eagerly.

Both of these studies explored the use of systemic tranexamic acid for treatment of PPH after the diagnosis has been made. However, no studies have explored the use of topical tranexamic acid given prophylactically to reduce bleeding in patients undergoing caesarean deliveries and to aid surgical haemostasis intra-operatively.

1.4 DOSE RATIONALE

The optimum dose of topical tranexamic acid required to reduce bleeding is not know. According to the Cochrane review on topical tranexamic acid, there was an overall 29% reduction of blood loss with topical tranexamic acid after analyzing 29 studies involving 2612 patients. The concentration of tranexamic acid used in these trials ranged from 0.7mg/ml to 100 mg/ml of saline solution.

The dose of topical tranexamic acid used in this study was selected based on the findings of a systemic review and meta-analysis on the use of topical tranexamic acid in total knee replacements which demonstrated that a dose >2g significantly reduces transfusion requirements. This is supported by a recent review of topical tranexamic acid in hip and knee arthroplasty in 2014 which suggest greater reductions in blood loss and transfusion with increasing dose. The investigators will be using 2g in 20mls solution of tranexamic acid diluted with 100mls of normal saline 0.9% yielding a concentration of 16.7mg/ml saline solution of topical tranexamic acid and it is postulated that this concentration of tranexamic acid should result in a 25% reduction in bleeding based on the existing clinical data.

1.5 OFF LABEL ROUTE OF ADMINISTRATION

Tranexamic acid is commonly prescribed in the oral or intravenous form. It has a good safety profile even when given systemically and the adverse effects related to the topical route are postulated to be less compared to the standard route of administration due to reduced systemic absorption of the drug. Furthermore, topical tranexamic acid is already used in clinical practice in many countries and there are many systematic reviews attesting to its efficacy and safety. Approval for the off-label route of administration of this drug has been obtained from the National Pharmaceutical Control Bureau and the Ministry of Health, Malaysia prior to the commencement of this trial.

1.6 POTENTIAL RISKS

Tranexamic acid has a well-documented safety profile. When given systemically (oral or intravenous) the adverse effects are as detailed in Table 1.

Table 1: Adverse Effects of Systemic Tranexamic Acid

Common (may affect up to 1 in 10 users) • Effects on the stomach and intestines: nausea, vomiting, diarrhoea (especially oral route)

Uncommon (may affect 1 to 10 in 1000 users)

• Effects on the skin: rash

Rare (frequency not known from available data)

* Effects on the haematological system: malaise with hypotension (especially if injected too quickly intravenously), arterial or venous thrombosis
* Effects on the nervous system: convulsions (in cases of misuse where high doses of intravenous tranexamic acid are given)
* Effects on the eyes: vision disturbances including impaired colour vision
* Effects on the immune system: allergic reactions

(For a more comprehensive list, please refer to the product information leaflets.)

The topical route of tranexamic acid is chosen as the investigators hypothesize that topical administration when compared to systemic routes would offer comparable clinical benefits in controlling bleeding but at the same time be safer in terms of causing potential adverse effects. The advantage of a more targeted action of the drug at the site of bleeding and reduced systemic absorption of topical tranexamic acid will mean that the adverse effects are likely be rare and those that are of relevance as listed as follows:

Table 2: Potential Adverse Effects of Topical Tranexamic Acid

* Effects on the haematological system: arterial or venous thrombosis
* Effects on the immune system: allergic reactions

Although tranexamic acid may theoretically increase the risk of thromboembolic events, systematic review of the drug in 2007 when given intravenously did not demonstrate any statistically significant increase in the risks of any thromboembolic events as showed in Table 3.

Table 3: Effects of Tranexamic Acid

Events Relative Risk (95% CI) Myocardial infarction 0.96 (0.48-1.90) Stroke 1.25 (0.47-3.31) Deep vein thrombosis 0.77 (0.37-1.61) Renal Failure 0.73 (0.16-3.32)

The investigators therefore concluded that topical tranexamic acid is likely to have minimal side effects on the study subjects.

1.7 POTENTIAL BENEFITS

Significant advantages of using topical tranexamic acid over systemic administration would include ease of use, targeted direct action of the drug at the site of bleeding with reduction in systemic complications, no risk of the drug entering the foetal circulation as the drug is administered only after delivery of the baby and placenta, and reduced adverse effects of the drug on the mother and the breast fed baby as the systemic absorption of the drug is unlikely to be significant. Ideally, we should also measure serum tranexamic acid and compare these to levels after systemic administration of the same dose of drug but this was not done due to limitation of cost and resources.

If found to be effective, the investigators' study has potential health benefits to mothers with moderate to high risks of bleeding in caesarean sections by reducing blood loss in surgery and also the complications associated with bleeding. The use of topical tranexamic acid can be incorporated into routine everyday use for these groups of patients and this practice can be easily implemented even in hospitals with limited resources, as it is simple, inexpensive and has minimal adverse effects. Reduced bleeding and better surgical haemostasis can also translate into shorter operating time, reduced risks of blood transfusion, better patient outcome and savings to the cost of healthcare.

1.8 SUBJECT RECRUITMENT AND SCREENING

Parturients planned for caesarean sections and who have increased risks of bleeding as stated in the inclusion criteria would be referred to the investigating team for screening. Subjects who fulfill all the inclusion and exclusion criteria and who consents to participate in the study after proper explanation would be recruited.

Written informed consent will be obtained from every patient prior to participation in this study. The investigator shall inform every subject in detail regarding the nature of this study, its purpose, the treatments and the probability of random assignment to the treatment groups, those aspects of the study that are experimental, the procedures involved, the possible risks, the reasonably expected benefits and the expected duration and the approximate number of subjects involved and their responsibilities. Consent will be obtained on a voluntary basis and refusal to participate in this study will not affect patient's subsequent medical treatment or relationship with the treating physicians.

Advance information will be provided where possible to parturients who are identified to be moderate to high risk for bleeding during their antenatal follow up. This includes a brief summary of the trial and the Patient Information Sheet, which will be made available at the antenatal clinic. All parturients planned for elective surgery will be recruited during their pre-operative assessment one day prior to the surgery.

Parturients planned for emergency surgery who fulfill the eligibility criteria for the study will be approached with the agreement of the obstetric team as soon as the decision of caesarean section is made. The Patient Information Sheet will be provided and the study will be discussed with her and an informed written consent will be obtained. Parturients with urgent indications for surgery where the timing of the caesarean section would be critical in determining the maternal and/or foetal outcomes will not be recruited as there would be insufficient time for them to give proper informed consent to participate in the study.

Patients who are deemed not competent to give proper consent as a result of altered state of mind due to existing illness, suffering from severe pain or side effects of drugs given will be excluded from the trial.

1.9 WITHDRAWAL OF SUBJECTS

Subjects may be withdrawn from the study by the study investigators prior to the expected completion of that subject if there are any safety concerns or failure of subject to adhere to protocol requirements which arises after recruitment process (e.g. disease progression, new contraindications to the use of tranexamic acid, or there is a change in the planned surgery where the patient may no longer fulfill the inclusion and exclusion criteria).

Patients enrolled in the trial may also withdraw their consent and discontinue their participation at any time without penalty or loss of benefits to which they are otherwise entitled to and their subsequent medical treatment or relationship with the treating physicians will not be affected. The study investigators would seek to document the reason(s) for subject consent withdrawal for documentation purposes unless the subject refuses to divulge their reason(s) for withdrawing from the study, whereby their decision would be respected.

In the event of subject consent withdrawal, the study investigator would clarify with the subject whether they wish to withdraw from all components of the trial or would they allow follow-up data collection activities to continue and the importance of obtaining follow-up safety data about the subject would be explained. All data already collected up to the point of subject withdrawal will be retained and analysed and attempts would also be made to obtain permission from the subjects who withdrew to record their follow-up safety data up to the end of subject follow-up period as described in the protocol.

1.10 METHODS OF RANDOMIZATION

Patients recruited into the trial will be randomized into 2 treatment groups; TXA group (Tranexamic acid 2g in 20mls solution diluted into 100mls of sterile sodium chloride 0.9% solution) or the Control group (120mls of sterile sodium chloride 0.9% solution) using software Research Randomizer (www.randomizer.org) and will be referred to as Group A and Group B respectively. This random assignment will be kept in sealed envelopes that will be marked with numbers corresponding to the sequence of patient's recruitment into the study.

1.11 STUDY PROCEDURES

1. The investigators will apply for special permission from the National Pharmaceutical Control Bureau and the Ministry of Health, Malaysia for the off-label route of administration of the tranexamic acid prior to the commencement of this trial.
2. Ethics approval will be obtained from the Malaysia Research Ethics Committee.
3. Patients who fulfill the inclusion and exclusion criteria will be recruited into the study.
4. Written informed consent will be obtained and patients will be randomized to 2 groups: The TXA group will receive 2g of topical tranexamic acid diluted in 100 ml of sodium chloride 0.9% during surgery whereas the Control group will receive 120ml of sodium chloride 0.9%.
5. Patients' risk factors for bleeding during caesarean sections will be assessed and documented.
6. The same surgical team will conduct the caesarean sections and they will carry out the surgery in a similar manner after patients are anaesthetised as per local practice. Only patients who received regional anaesthesia will be included in the study. Patients who are planned for general anaesthesia will not be recruited and those who required conversion to general anaesthesia after recruitment due to various reasons (i.e. failed regional anaesthesia, prolonged operation, maternal request) prior to administration if the study therapy will be drop out from the study and the reason for dropping out should be clearly documented in the case report form (CRF).
7. The study therapy will be administered only after the delivery of the baby and the placenta. The attending surgeon should first attempt to secure the initial haemostasis by applying clamps at both ends of the surgical incision on the uterus. The placenta should be removed completely and two pieces of gauze used to thoroughly evacuate any remnants of conception from the upper and lower segment of the uterus (above and below the incision site) to ensure no remnants are sticking to the placental bed. The solution containing the study drug should then be syringed out from the gallipot using a sterile 20ml syringe. 60mls of the solution will be applied topically to the placental bed as identified by the surgeon carrying out the surgery by spraying the solution into the cavity over the placental bed. Another 30mls of the solution will be applied to the open incision wound. The surgeon will then proceed to close the first layer of the uterus in the usual manner. After closure of the first layer, the repaired incision will then be dried with an abdominal pack. Any active spurting vessels will be secured prior to applying the remaining sample of study drug solution. Once the surgeon is satisfied there are no active vessel bleeders, another 30mls of the study drug solution is then applied topically on the closed incision wound in a similar manner. The rest of surgery is then carried out as per routine practice.
8. At the end of the surgery, intra-operative blood loss will be documented by the circulating nurse and the anaesthetist in charge. Blood loss from the suction bottles is measured and all gauzes and drapes soaked with blood will be weighed using a sensitive weighing scale (up to 0.01g accuracy) and the total blood loss is documented in the CRF. Care is taken to separate amniotic fluids loss and actual blood loss by using different suction catheters during the operation.
9. Intra-operative blood loss will be calculated using the following formula:

   Total intra-operative blood loss (mls) = i. Blood volume measured in suction bottle ii. Plus (+) wet weight of all gauzes and drapes soaked with blood iii. Minus (-) dry weight of all gauzes and drapes soaked with blood (Assumption of 1 gram of blood is equivalent to 1 ml of blood)
10. Haematocrit levels are monitored at baseline (prior to caesarean section) and at 6 hours post-operatively.
11. Subjects who have haemoglobin less than 70g/dl or have clinical symptoms of anemia will be transfused. All blood products transfused intra-operatively and in the first 24 hours after surgery will be documented.
12. Use of additional uterotonics in addition to the routine 5 units oxytocin bolus at delivery of the baby and the subsequent maintenance of 40 units oxytocin over 6 hours will be documented in the CRF.
13. Patients who has massive haemorrhage and who may benefit from the use of systemic antifibrinolytics based on the judgement of the attending physician can be given tranexamic acid intravenously or other antifibrinolytics according to clinical requirements and the types of drug and dosage given should be documented in the CRF.
14. Patients are followed up till the time of discharge and the length of stay in hospital will be compared. Complications rate (number of events) post caesarean section as a result of bleeding (i.e. relaparotomy, hysterectomy, internal iliac artery ligations, embolization) and mortality will also be compared in both groups of patients.
15. Serious adverse events (SAR) potentially related to the use of topical tranexamic acid (e.g. allergic reactions and thrombotic events including myocardial infarction, strokes, pulmonary embolism, deep vein thrombosis) will be monitored closely by the attending physician up to the time of discharge. The principal investigator will be informed immediately of such events and the patient will be referred to the medical and intensive care unit for further management. A report regarding the SAR will be submitted to the relevant authorities.
16. Subjects will be followed up to 30 days post caesarean section through telephone or email after discharge from hospital and any adverse events made known to the investigators by the patient or the primary team will be documented in the CRF.

1.12 STATISTICAL PLAN

Sample size calculation was done using the Power and Sample Size Calculation Version 3.0 January 2009.

The average blood loss expected in a lower segment caesarean section is estimated to be around 600 ± 187ml.5 A 25 % reduction in blood loss is predicted with the use of topical tranexamic acid. A sample size of 36 patients per arm would be required in this study assuming a power of 90 percent and a significant level of 0.05. A 20 percent drop out rate is projected, therefore a total of 84 patients will be enrolled with 42 patients in each arm of the study.

All data will be collected into the CRF. The data will be keyed in using the Statistical Package for the Social Sciences (SPSS) Program for Windows Version 19. All dosed subjects will be included in data analysis. Data collected will be assessed further for their distribution. Continuous, numerical and parametric data (e.g. total blood loss measured, haematocrit trends in both groups) will be analysed using independent student t-test. Non-parametric numerical data will be analysed using the Mann Whitney-U test where else categorical data collected will be tested using the Chi-square test (e.g. risk factors for bleeding, transfusion requirements) as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Parturients aged more than 18 years old
2. American Society of Anesthesiologists (ASA) physical status class 1 to 3
3. Parturients planned for caesarean sections (both emergency and elective) under regional anaesthesia
4. Parturients who have increased risks of bleeding during caesarean deliveries as follows:

Moderate Risk for Bleeding

* Induction of labour
* Prolonged labour >12 hours
* Large baby > 4kg
* Pyrexia in labour
* Age > 40 years (not multiparous)
* Obesity (BMI >35)
* Anaemia (Hb < 9g/dl)
* Multigravida
* Previous history of PPH
* Previous scars

High Risk for Bleeding

* Known bleeding disorders (congenital or acquired)
* Multiple pregnancies
* Preeclampsia and pregnancy induced hypertension
* Placenta praevia
* Placenta accreta/increta/percreta
* Placenta abruption

Exclusion Criteria:

1. Parturients who have an urgent/emergency indication for caesarean sections where timing of the operation may be critical in determining the maternal and/or foetal outcomes
2. Patients who are planned for caesarean sections under general anaesthesia
3. Patients who are already clinically bleeding prior to surgery
4. Parturients who received blood transfusion within 48 hours prior to the caesarean section
5. Patients with known allergy to tranexamic acid
6. Patients with clear contraindications for tranexamic acid (e.g. thromboembolic event, history of convulsions)
7. Patients with severe renal failure with creatinine clearance <10

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Total intra-operative blood loss in the Tranexamic Acid (TXA) group compared to the Control group | From the start of the surgery (first surgical incision) up to the end of the surgery (at wound closure)
  Total intra-operative blood loss will be measured at the end of the surgery (at wound closure).
  The following formula will be used:
  Total intra-operative blood loss (ml) = A + B - C where A = Blood volume in suction bottle (ml) B = Wet weight of all gauzes and drapes soaked with blood (g) C = Dry weight of all gauzes and drapes soaked with blood (g) (assumption of 1 gram of blood is equivalent to 1ml of blood) The blood loss quantified will be documented in subjects case report form

SECONDARY OUTCOMES:
Transfusion requirements in terms of number of red blood cell packets transfused up to 24 hours post surgery | From start of surgery (first surgical incision) up to 24 hours post surgery (wound closure)
  The number of red blood cell packets (number of pints) transfused in all patients from the start of the surgery up to 24 hours post surgery will be documented in each subject's case report form and the transfusion requirements will be compared between both groups.
Haematocrit trends at baseline (Pre-operative) and at 6 hours post surgery in the TXA group and the Control group | Pre-operatively within 24 hours prior to start of surgery (before surgical incision) up to 6 hours from the end of surgery (wound closure)
  Subjects full blood count will be taken pre-operatively within 24 hours prior to start of surgery (baseline) and at 6 hours from the end of the surgery (wound closure) to measure the haematocrit trends in both study groups and these values will be documented in the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Li Lee, FANZCA, Principal Investigator — Department of Anaesthesia, Hospital Tengku Ampuan Rahimah, Ministry of Health, Malaysia
Locations (1):
- Hospital Tengku Ampuan Rahimah, Klang, Selangor, Malaysia

REFERENCES:
- [Background] AbouZahr C. Global burden of maternal death and disability. Br Med Bull. 2003;67:1-11. doi: 10.1093/bmb/ldg015. PMID 14711750
- [Background] Al Kadri HM, Al Anazi BK, Tamim HM. Visual estimation versus gravimetric measurement of postpartum blood loss: a prospective cohort study. Arch Gynecol Obstet. 2011 Jun;283(6):1207-13. doi: 10.1007/s00404-010-1522-1. Epub 2010 May 28. PMID 20508942
- [Background] Larsson C, Saltvedt S, Wiklund I, Pahlen S, Andolf E. Estimation of blood loss after cesarean section and vaginal delivery has low validity with a tendency to exaggeration. Acta Obstet Gynecol Scand. 2006;85(12):1448-52. doi: 10.1080/00016340600985032. PMID 17260220
- [Background] Knight M, Callaghan WM, Berg C, Alexander S, Bouvier-Colle MH, Ford JB, Joseph KS, Lewis G, Liston RM, Roberts CL, Oats J, Walker J. Trends in postpartum hemorrhage in high resource countries: a review and recommendations from the International Postpartum Hemorrhage Collaborative Group. BMC Pregnancy Childbirth. 2009 Nov 27;9:55. doi: 10.1186/1471-2393-9-55. PMID 19943928
- [Background] Ortmann E, Besser MW, Klein AA. Antifibrinolytic agents in current anaesthetic practice. Br J Anaesth. 2013 Oct;111(4):549-63. doi: 10.1093/bja/aet154. Epub 2013 May 9. PMID 23661406
- [Background] Coats T, Roberts I, Shakur H. Antifibrinolytic drugs for acute traumatic injury. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD004896. doi: 10.1002/14651858.CD004896.pub2. PMID 15495129
- [Background] Adler Ma SC, Brindle W, Burton G, Gallacher S, Hong FC, Manelius I, Smith A, Ho W, Alston RP, Bhattacharya K. Tranexamic acid is associated with less blood transfusion in off-pump coronary artery bypass graft surgery: a systematic review and meta-analysis. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):26-35. doi: 10.1053/j.jvca.2010.08.012. Epub 2010 Nov 5. PMID 21115366
- [Background] Tzortzopoulou A, Cepeda MS, Schumann R, Carr DB. Antifibrinolytic agents for reducing blood loss in scoliosis surgery in children. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD006883. doi: 10.1002/14651858.CD006883.pub2. PMID 18646174
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Novikova N, Hofmeyr GJ. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007872. doi: 10.1002/14651858.CD007872.pub2. PMID 20614466
- [Background] Ducloy-Bouthors AS, Jude B, Duhamel A, Broisin F, Huissoud C, Keita-Meyer H, Mandelbrot L, Tillouche N, Fontaine S, Le Goueff F, Depret-Mosser S, Vallet B; EXADELI Study Group; Susen S. High-dose tranexamic acid reduces blood loss in postpartum haemorrhage. Crit Care. 2011;15(2):R117. doi: 10.1186/cc10143. Epub 2011 Apr 15. PMID 21496253
- [Background] Shakur H, Elbourne D, Gulmezoglu M, Alfirevic Z, Ronsmans C, Allen E, Roberts I. The WOMAN Trial (World Maternal Antifibrinolytic Trial): tranexamic acid for the treatment of postpartum haemorrhage: an international randomised, double blind placebo controlled trial. Trials. 2010 Apr 16;11:40. doi: 10.1186/1745-6215-11-40. PMID 20398351
- [Background] Panteli M, Papakostidis C, Dahabreh Z, Giannoudis PV. Topical tranexamic acid in total knee replacement: a systematic review and meta-analysis. Knee. 2013 Oct;20(5):300-9. doi: 10.1016/j.knee.2013.05.014. Epub 2013 Jun 28. PMID 23815893
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760
- [Background] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Background] Alshryda S, Sukeik M, Sarda P, Blenkinsopp J, Haddad FS, Mason JM. A systematic review and meta-analysis of the topical administration of tranexamic acid in total hip and knee replacement. Bone Joint J. 2014 Aug;96-B(8):1005-15. doi: 10.1302/0301-620X.96B8.33745. PMID 25086114
- See also: The Millennium Developmental Goals Report 2008 — http://www.un.org/millenniumgoals/2008highlevel/pdf/newsroom/mdg%20reports/MDG_Report_2008_ENGLISH.pdf
- See also: Postpartum Haemorrhage, Prevention and Management (Green-top Guideline No. 52) — https://www.rcog.org.uk/en/guidelines-research-services/guidelines/gtg52/